CLINICAL TRIAL: NCT03089385
Title: Development, Validation, and Implementation of a Clinical Decision Tool for Blood Pressure Management in Patients on Hemodialysis
Brief Title: Use of a Hypertension Tool to Manage Blood Pressure in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-9951
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation group (Experimental): This group will have the hypertension tool implemented on them.
  Interventions: Other: Hypertension tool
- Control group (No Intervention): This group will not have the tool implemented.

INTERVENTIONS:
Other: Hypertension tool — An algorithm developed by staff at UHN to help manage hypertension in hemodialysis patients.
  Arms: Implementation group

SUMMARY:
The objective of this project is to develop, validate, and implement a tool to help manager hypertension in patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Receiving in-centre HD for at least 3 months
* Considered hypertensive based on a median intradialytic blood pressure ≥ 140/90 mmgHG

Exclusion Criteria:

* Are unable to provide informed consent
* Are deemed medically unstable by the primary physician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Battistella, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada